CLINICAL TRIAL: NCT03478059
Title: Exploring the Role of Combined Cognitive and Motor Dual-task Assessment and Rehabilitation for Individuals With Residual Symptoms After mTBI
Brief Title: Dual-task Assessment and Rehabilitation for Individuals With Residual Symptoms After mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Margaret Weightman, Senior Scientific Advisor, Allina Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKMW-1701
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Brain Injury Traumatic Mild; Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Traumatic Brain Injury (Experimental): 60 minute, 3 times per week, 6 week long Cognitive and Motor Dual-task Intervention program. The intervention will consist of 6 stations that target known motor and cognitive impairments after mTBI.
  Subjects with mTBI residuals will be gently progressed through exercise stations in an individually tailored fashion.
  Interventions: Behavioral: Cognitive and Motor Dual-task Intervention
- Healthy Control (Other): 60 minute, 3 times per week, 6 week long Cognitive and Motor Dual-task Intervention program. The intervention will consist of 6 stations that target known motor and cognitive impairments after mTBI.
  In addition to providing comparison data, the healthy control, athletic 18-34 year old subjects will be used to identify levels and intensity of progressions of dual-task training stations appropriate for highly trained athletes and military personnel recovering from concussion.
  Interventions: Behavioral: Cognitive and Motor Dual-task Intervention

INTERVENTIONS:
Behavioral: Cognitive and Motor Dual-task Intervention — The intervention will take place 3 times per week for 6 weeks (60 minutes/session) and employs motor and cognitive challenges. It is based on known motor and cognitive deficits after mTBI and is structured using a theoretical framework published in another domain of neurologic disease. The intervention will consist of 6 stations that target known motor and cognitive impairments after mTBI. Each station will have 3 levels of difficulty with optional cognitive progressions. Subjects will spend 8 minutes at each station with a 2 minute transition/rest period between stations and will be progressed in motor and cognitive difficulty as able.

SUMMARY:
This research aims to develop an intervention that combines mTBI-specific motor and cognitive challenges into a progressive and challenging rehabilitation program. We plan to develop and refine a combined motor and cognitive intervention using healthy athletic young adults (n=12) and people with a positive history of non-resolving mTBI (n=12). We will conduct limited feasibility testing by conducting 6 week training sessions with each subject group. We also plan to identify best measures for determining readiness for duty or full function by incorporating and testing 3 dual-task assessment measures using state-of-the-art wearable sensors to quantify movement.

ELIGIBILITY:
Inclusion criteria-healthy control:

* Adults aged 18-34 years of age.
* Strong history of athletic participation including high school and collegiate varsity and/or club sports
* Current sport or recreational sport participation at least 3 days per week
* Willingness to participate in 3 times a week 60 minute exercise program conducted at Courage Kenny Research Center (CKRC).

Exclusion Criteria-healthy control:

* History of concussion.
* History of orthopedic or neurologic diagnosis (stroke, multiple sclerosis, Parkinson's Disease, etc.) interfering with subject's ability to exercise
* Unwilling to exercise.
* At risk for cardiopulmonary disease as defined by the American College of Sports Medicine.
* Active medical contraindications by self-report after explanation of dual-task exercise program.
* Active chemical dependency or major psychiatric disorders (ie., schizophrenia, major psychosis) by self-report.

Inclusion criteria-subjects with mTBI residual symptoms:

* Adults aged 18-50 years of age.
* Self-report of some consistent exercise or activity a minimum of 2-3 days per week.
* 3 weeks to 24 months post most recent concussion seeking treatment at Courage Kenny Rehabilitation Institute (CKRI) clinics
* Willingness to participate in 3 times a week 60 minute exercise program conducted at CKRC.

Exclusion Criteria- subjects with mTBI residual symptoms:

* History of orthopedic or neurologic diagnosis (stroke, multiple sclerosis, Parkinson Disease, etc.) interfering with subject's ability to exercise
* Unwilling to exercise.
* At risk for cardiopulmonary disease as defined by the American College of Sports Medicine.
* Active medical contraindications by self-report after explanation of dual-task exercise program,
* Active chemical dependency or major psychiatric disorders (ie., schizophrenia, major psychosis).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in peak velocity turns during Instrumented Stand and Walk Test | At baseline and after 6 weeks of intervention
  Change in peak velocity during 180 degree turns during Instrumented Stand and Walk Test in single task (ST) and dual-task (DT) conditions. DT condition involves grid memorization task.

SECONDARY OUTCOMES:
Change in peak turning velocity during walking a custom turning course | At baseline and after 6 weeks of intervention
  Change in peak turning velocity during walking a custom turning course in ST and DT conditions.
Change in peak turning velocity during running an agility course | At baseline and after 6 weeks of intervention
  Change in peak turning velocity during running an agility course in ST and DT conditions.
Change in medial -lateral (coronal plane) sway area during eyes closed, narrowed stance | At baseline and after 6 weeks of intervention
  Change in medial -lateral (coronal plane) sway area during eyes closed, narrowed stance in ST and DT conditions.
Change in Beck Depression Inventory-II | At baseline and after 6 weeks of intervention
  Change in Beck Depression Inventory-II: 21 item self-administered questionnaire that measures intensity of depression.
Change in Beck Anxiety Inventory | At baseline and after 6 weeks of intervention
  Change in Beck Anxiety Inventory: 21 item self-administered questionnaire measuring subjective, somatic, or panic-related symptoms of anxiety.
Change in Patient-specific Functional Scale | At baseline and after 6 weeks of intervention
  Change in Patient-specific Functional Scale -quantifies the amount of functional limitation secondary to symptoms in up to 3 activities that are relevant to the individual patient. 0 to 10 scale, where 0 = unable to perform activity and 10 = able to perform activity at same level as before injury or problem.
Change in Neurobehavioral Symptom Inventory (NSI) | At baseline and after 6 weeks of intervention
  Change in Neurobehavioral Symptom Inventory (NSI): Self-report of residual symptoms "in last 2 weeks", a measure of post-TBI symptom severity, 0-4 scale on 22 symptom questions.
Rey Auditory Verbal Learning Test Score | At baseline
  Rey Auditory Verbal Learning Test which measures verbal learning and memory (short-term)
Comprehensive Trails Making Test Score | Baseline
  Comprehensive Trails Making Test which measures set shifting, attention, psychomotor speed
Verbal Fluency Test Score | Baseline
  Verbal Fluency which tests verbal ability and executive control
NAB Digits Forward/Digits Backward Test Score | Baseline
  NAB Digits Forward/Digits Backward Test which measures attentional capacity and auditory working memory
Stroop Color-Word Test Score | Baseline
  Stroop Color-Word Test to evaluate sustained and selective attention as well as freedom from distractibility and inhibitory control.
Wide Range Achievement Test-4 Reading Score | Baseline
  Wide Range Achievement Test-4 Reading will be used as an estimate of premorbid intellect

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Weightman, PT, PhD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States